CLINICAL TRIAL: NCT06514703
Title: Comparative Study of CT and Fluoroscopic Guided Genicular Nerve Ablation in the Treatment of Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Awad Bessar, Assistant Professor of Diagnostic and Interventional Radiology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTFGNA-KOA
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Osteoarthritis; Genicular Nerve Ablation; CT-guided Ablation; Fluoroscopic-guided Ablation; Pain Management; Minimally Invasive Procedures; Patient Satisfaction
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this randomized controlled trial, a partial blinding strategy is employed where only the outcomes assessors are blinded to intervention group assignments. Given the distinct nature of the CT-guided and fluoroscopic-guided procedures, it is impractical to blind participants and care providers. Operators performing the ablation and participants will be aware of the imaging technique used. However, to ensure unbiased evaluation of clinical outcomes, outcomes assessors will not know participants' group assignments. This measure is crucial for preventing observer bias in assessing primary and secondary outcomes such as pain relief, functional improvement, and patient satisfaction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT-Guided Genicular Nerve Ablation (Experimental): Participants in this arm will undergo genicular nerve ablation using computed tomography (CT) guidance. The procedure involves precise needle placement based on CT imaging to effectively target the genicular nerves responsible for transmitting pain signals from the knee.
  Interventions: Procedure: CT-Guided Genicular Nerve Ablation
- Fluoroscopic-Guided Genicular Nerve Ablation (Active Comparator): Participants in this arm will receive genicular nerve ablation using fluoroscopic guidance. The procedure utilizes real-time fluoroscopy to guide needle placement for the ablation of the genicular nerves.
  Interventions: Procedure: Fluoroscopic-Guided Genicular Nerve Ablation

INTERVENTIONS:
Procedure: CT-Guided Genicular Nerve Ablation — This procedure involves using computed tomography (CT) imaging to guide the precise placement of a needle for the ablation of genicular nerves in the knee. The goal is to disrupt the pain signals caused by osteoarthritis, providing long-term pain relief. The intervention is performed under local anesthesia and is aimed at patients who have not responded adequately to conservative pain management strategies.
  Arms: CT-Guided Genicular Nerve Ablation
Procedure: Fluoroscopic-Guided Genicular Nerve Ablation — This procedure utilizes fluoroscopy to accurately guide the needle placement for the ablation of genicular nerves associated with osteoarthritis knee pain. The technique focuses on minimizing pain and improving functional mobility by disrupting nerve pathways that transmit pain signals. Like the CT-guided approach, it is intended for use in patients whose symptoms have not been sufficiently managed with non-invasive treatments.
  Arms: Fluoroscopic-Guided Genicular Nerve Ablation

SUMMARY:
The goal of this study is to evaluate the comparative effectiveness of CT-guided and fluoroscopic-guided genicular nerve ablation in reducing knee pain and improving function in adults diagnosed with knee osteoarthritis refractory to conservative treatment.

The main questions it aims to answer are:

* Does CT-guided genicular nerve ablation provide superior pain relief compared to fluoroscopic-guided genicular nerve ablation?
* Is there a significant difference in functional improvement between the two techniques?

Researchers will compare the outcomes between the CT-guided and fluoroscopic-guided groups to determine which method achieves better pain relief, functional enhancement, safety profile, and patient satisfaction.

Participants will:

* Undergo either CT-guided or fluoroscopic-guided genicular nerve ablation.
* Attend scheduled follow-up visits to assess pain levels, knee function, and any adverse events.
* Complete standardized questionnaires to provide feedback on pain relief, functional improvement, and overall satisfaction with the procedure.

DETAILED DESCRIPTION:
Background:

Knee osteoarthritis is a chronic degenerative joint disease affecting millions worldwide, characterized by progressive cartilage loss, inflammation, and pain. Despite various treatment options such as intra-articular corticosteroids, viscosupplementation, and PRP injections, many patients experience inadequate relief or adverse effects. Genicular nerve ablation has emerged as a promising minimally invasive technique to alleviate chronic knee pain by interrupting pain transmission from the genicular nerves to the central nervous system.

Rationale:

The rationale for comparing CT-guided and fluoroscopic-guided genicular nerve ablation lies in optimizing treatment outcomes while ensuring patient safety and satisfaction. CT-guided procedures offer unparalleled precision in nerve localization, potentially enhancing the accuracy of nerve ablation and improving clinical outcomes. However, this method involves higher radiation exposure compared to fluoroscopic guidance, which utilizes real-time imaging with lower radiation doses. Understanding which approach provides superior pain relief, functional improvement, and patient satisfaction is crucial for optimizing treatment protocols and guiding clinical practice.

Objectives:

Primary Objective:

1) Evaluate the efficacy of CT-guided and fluoroscopic-guided genicular nerve ablation in reducing knee pain, as measured by the visual analog scale (VAS), at 3 months post-procedure.

Secondary Objectives:

1. Evaluate changes in knee function using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), a validated scoring system specifically designed for osteoarthritis.
2. Monitor and document any procedure-related adverse events to compare the safety profiles of both techniques.
3. Evaluate patient satisfaction using the structured Patient Satisfaction Questionnaire (PSQ)

Study Design:

This study is a randomized controlled trial (RCT) aimed at evaluating the comparative effectiveness of CT-guided versus fluoroscopic-guided genicular nerve ablation. Eligible patients will be randomly allocated to one of the two treatment groups. Given the specific nature of the interventions, it may not be possible to blind participants or operators; however, to minimize potential bias, outcome assessors will be blinded to the treatment assignments.

Participants:

* Inclusion Criteria: Adults aged 45-80 diagnosed with knee osteoarthritis refractory to conservative treatment, characterized by persistent knee pain despite medication and physical therapy.
* Exclusion Criteria: Patients with contraindications to genicular nerve ablation procedures (e.g., allergy to local anesthetics, active infection at the procedure site), or recent knee surgery within the last six months.

Interventions:

1. CT-guided Genicular Nerve Ablation: Patients will undergo CT-guided genicular nerve ablation, involving meticulous planning of needle placement under CT imaging to accurately target the genicular nerves responsible for knee pain. Ablation parameters will be standardized to ensure consistency across procedures.
2. Fluoroscopic-guided Genicular Nerve Ablation: Patients assigned to this group will undergo genicular nerve ablation under fluoroscopic guidance, utilizing real-time X-ray imaging to guide needle placement and confirm adequate nerve coverage before ablation.

Outcomes:

* Primary Outcome: Reduction in knee pain measured by visual analog scale (VAS) at 3 months post-procedure.
* Secondary Outcomes
* Improvement in knee function measured by changes in WOMAC scores over the follow-up period.
* Incidence and nature of any procedure-related adverse events
* Patient-reported outcomes regarding satisfaction, using the structured PSQ

Follow-Up:

Participants will be closely monitored post-procedure with scheduled follow-up visits at 1 week, 1 month, 3 months, and 6 months. These visits will include clinical assessments, pain evaluations, functional tests, and documentation of any adverse events.

Conclusion:

This study aims to provide valuable insights into the comparative effectiveness, safety, and patient satisfaction of CT-guided versus fluoroscopic-guided genicular nerve ablation in the management of knee osteoarthritis. By rigorously evaluating these techniques, the findings will inform clinical decision-making, optimize treatment strategies, and pave the way for future research aimed at enhancing outcomes for patients suffering from chronic knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45 to 80 years.
* Diagnosed with knee osteoarthritis.
* Knee osteoarthritis refractory to conservative treatment.
* Able to provide informed consent.
* Agree to follow the study procedures and attend follow-up visits.

Exclusion Criteria:

* Prior knee surgery within the last six months.
* Contraindications to genicular nerve ablation (e.g., certain types of infections, bleeding disorders).
* Severe comorbid conditions that may interfere with the study outcomes (e.g., rheumatoid arthritis, other severe autoimmune diseases).
* Current participation in another clinical trial that could interfere with the outcomes of this study.
* Allergy or sensitivity to the materials used in the ablation procedures.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Knee Pain | 3 months post-procedure
  This measure assesses the change in knee pain as reported by participants using the Visual Analog Scale (VAS). A lower score indicates less pain, signifying an improvement.

SECONDARY OUTCOMES:
Improvement in Knee Function | Assessed at baseline, 1 month, 3 months, and 6 months post-procedure
  Assessed by changes in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores, which measure pain, stiffness, and physical function of the knee and hip joints. A lower WOMAC score indicates better joint function.
Incidence of Procedure-Related Adverse Events | From the time of procedure up to 6 months
  Monitoring and recording any adverse events related to the genicular nerve ablation procedures
Patient Satisfaction with the Procedure | 3 months post-procedure
  Measured using a structured patient satisfaction questionnaire (PSQ) to gauge participants' satisfaction with the pain relief and overall experience of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Bessar, MD, PhD, Principal Investigator — Assistant Professor of Diagnostic and Interventional Radiology, Zagazig Uni.
Locations (1):
- Zagazig University, Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) with other researchers. This decision is based on considerations related to patient confidentiality, data privacy concerns, and the absence of a current infrastructure for secure data sharing. The primary results of the study will be published in peer-reviewed journals and presented at scientific conferences, ensuring that the findings are accessible to the broader research community.